CLINICAL TRIAL: NCT07301970
Title: Population Pharmacokinetics of Remifentanil for Analgesia and Sedation in Low-Weight Critically Ill Patients Receiving Mechanical Ventilation
Brief Title: Population Pharmacokinetics of Remifentanil in Low-Weight Critically Ill Patients
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiang Li, Director, Shanghai Minhang Central Hospital
Other Study IDs: 2025-007-01K
Record Dates: First submitted 2025-11-29; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-09

CONDITIONS: Critical Illness; Pain
MeSH Terms: conditions — Critical Illness; Pain | interventions — Remifentanil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low-weight group: BMI < 18.5
  Interventions: Drug: Remifentanil
- Normal-weight group: 18.5 ≤ BMI< 24
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Patients receive remifentanil for analgesia and sedation during mechanical ventilation. The administration follows standard ICU clinical practice, typically initiated at a continuous infusion rate (e.g., approximately 0.18 mg/h or weight-based equivalent) and titrated based on patient response.

SUMMARY:
The goal of this prospective clinical study is to learn about the population pharmacokinetics (PopPK), safety, and efficacy of remifentanil in low-body-weight patients in the Intensive Care Unit (ICU) who require mechanical ventilation. The main questions it aims to answer are:

1. What are the pharmacokinetic characteristics of remifentanil in low-weight ICU patients?
2. How does remifentanil (and concurrent propofol use) affect hemodynamic stability (such as blood pressure) and sedation efficacy in this population?

Participants receiving mechanical ventilation will receive remifentanil for analgesia and sedation according to a standardized protocol. They will undergo arterial blood sampling at specific time points to measure drug concentrations. Researchers will also record hemodynamic parameters. Additionally, a subset of patients receiving propofol as a rescue sedative will have plasma propofol concentrations measured to evaluate its influence on blood pressure changes.

DETAILED DESCRIPTION:
1. Background: Remifentanil is a lipophilic μ-opioid receptor agonist characterized by rapid onset and offset, making it ideal for analgosedation in the Intensive Care Unit (ICU). Body weight is a significant factor affecting its pharmacokinetics (PK). Low-body-weight patients may require different dosing strategies. This study aims to establish a population pharmacokinetic (PopPK) model for remifentanil in mechanically ventilated patients with low body weight and to evaluate its safety and efficacy, with a specific focus on hemodynamic stability.
2. Study Protocol & Dosing Strategy: This is a single-center, prospective observational study designed to reflect real-world clinical practice. Eligible patients requiring invasive mechanical ventilation will receive remifentanil for analgesia and sedation.

   * Co-administration: In accordance with standard ICU practice, remifentanil is often administered concurrently with propofol to ensure adequate sedation and analgesia.
   * Dosing Regimen: The administration of a loading dose is discretionary based on the patient's clinical condition; in many cases, a continuous infusion is initiated directly without a loading dose to maintain hemodynamic stability.
   * Infusion Rate: The continuous infusion is typically initiated at a standardized clinical rate (e.g., approximately 0.18 mg/h) or a weight-based equivalent.
   * Titration: Subsequent dosing is titrated dynamically based on clinical response (e.g., patient comfort, ventilator synchrony) and hemodynamic tolerance.
3. Pharmacokinetic Sampling (Sparse & Opportunistic): Blood samples are not collected at rigid clock times but are distributed to capture key PK phases:

   * Absorption/Distribution Phase: Samples collected within the first hour of infusion (e.g., 1-2 samples).
   * Steady State: Samples collected during stable continuous infusion.
   * Elimination Phase: Samples collected immediately prior to stopping the infusion and at multiple intervals after discontinuation.

5.Hemodynamic Assessment & Propofol Co-variate Analysis: Hemodynamic parameters (MAP, HR) are continuously monitored. Given that propofol is co-administered in most patients and significantly impacts hemodynamics, plasma propofol concentrations will be measured in a subset of patients. These data will be incorporated into the PopPK/PD analysis as a covariate to distinguish the hemodynamic effects of remifentanil from those of propofol.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old, regardless of sex;
* Normal weight: 18.5 kg/m² ≤ Body Mass Index (BMI) < 24 kg/m² or Low weight: BMI < 18.5 kg/m²;
* Admitted to the intensive care unit (ICU);
* Required invasive mechanical ventilation for more than 10 hours;
* The subject or their legal guardian has fully understood the potential risks and benefits of participating in this study and has signed the informed consent form.

Exclusion Criteria:

* Pregnant women;
* Presence of severe respiratory impairment or respiratory depression during the screening period;
* Known hypersensitivity to remifentanil or any of the excipients;
* Meeting other contraindications for opioid use

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients admitted to the Intensive Care Unit (ICU) requiring invasive mechanical ventilation who receive remifentanil for analgesia and sedation. The study population comprises two cohorts stratified by Body Mass Index (BMI): a low-body-weight group (BMI < 18.5 kg/m²) and a normal-body-weight control group (18.5 kg/m² ≤ BMI < 24 kg/m²).
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentration of Remifentanil | From the start of remifentanil administration, through the maintenance infusion phase, up to 2 hours after the end of infusion.
  Peripheral arterial blood samples (1mL each) drawn from an existing indwelling arterial blood pressure (ABP) catheter will be collected to determine the plasma concentration of remifentanil (unit: ng/mL). A sparse and opportunistic sampling strategy is employed to capture the full pharmacokinetic profile. Sampling points typically include:
  1. Absorption/Distribution Phase: Approximately 2 samples within the first 2 hours of administration;
  2. Maintenance Phase: Samples collected during steady-state infusion, and following dose adjustments to capture the new steady state (typically after re-equilibration);
  3. Elimination Phase: Approximately 3 samples within 2 hours after the end of infusion.

SECONDARY OUTCOMES:
Mean Arterial Pressure (MAP) | From baseline throughout the duration of drug infusion (up to approximately 48 hours).
  Evaluation of hemodynamic stability by measuring the absolute value of MAP. Reported in mmHg.
Plasma Concentration of Propofol | From the start of its administration, through the maintenance infusion phase, up to 2 hours after the end of infusion.
  Plasma propofol concentrations will be measured in the subset of patients who receive propofol as a rescue sedative or co-medication. This data will be used as a covariate in the PK/PD analysis to differentiate the hemodynamic effects of propofol from those of remifentanil.
Heart Rate | From baseline throughout the duration of drug infusion (up to approximately 48 hours).
  Evaluation of hemodynamic stability by measuring Heart Rate. Reported in beats per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Li, Principal Investigator — Shanghai Minhang Central Hospital
Locations (1):
- Shanghai Minhang Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy restrictions and ethical considerations.